CLINICAL TRIAL: NCT01903109
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalence Study of Cevimeline 30 mg Capsules Under Fed Conditions
Brief Title: Crossover Bioequivalence Study of Cevimeline 30 mg Capsules Under Fed Conditions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CEVI-C30-PVFD-1
Record Dates: First submitted 2013-07-12; First posted 2013-07-19 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Dry Mouth
MeSH Terms: conditions — Xerostomia | interventions — cevimeline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cevimeline first, the Evoxac (Active Comparator): Single dose 30 mg cevimeline capsule, then single dose 30 mg Evoxac capsule (after washout period)
  Interventions: Drug: Cevimeline
- First Evoxac, then cevimeline (Active Comparator): Single dose 30 mg Evoxac capsule, then single dose 30 mg cevimeline capsule (after washout period)
  Interventions: Drug: Cevimeline

INTERVENTIONS:
Drug: Cevimeline
  Other Names: Evoxac

SUMMARY:
The objective of this study was to prove the bioequivalence of Roxane Laboratories' Cevimeline 30 mg under fed conditions

ELIGIBILITY:
Inclusion Criteria:

- No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to cevimeline or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 33 Days

CONTACTS AND LOCATIONS:
Overall Officials: Darin Brimhall, DO, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Las Vegas, Nevada, United States